CLINICAL TRIAL: NCT03731065
Title: Examining Exogenous Carbohydrate Oxidation From Glucose, Multiple Transportable Carbohydrates and Hydrogel Carbohydrate Drinks During Endurance Running
Brief Title: Exogenous Oxidation of Fructose-glucose Mixtures During Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Associate Professor, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MSES 17/18-001
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fructose-maltodextrin ingestion (Active Comparator): Ingestion of fructose and maltodextrin (glucose polymers) at a rate of 90 g carbohydrate per hour during two hours of treadmill running at 60%VO2peak.
  Interventions: Dietary Supplement: Fructose-maltodextrin
- Fructose-maltodextrin hydrogel ingestion (Experimental): Ingestion of fructose and maltodextrin (glucose polymers) encapsulated in alginate-pectin hydrogel, drinks at a rate of 90 g carbohydrate per hour during two hours of treadmill running at 60%VO2peak.
  Interventions: Dietary Supplement: Fructose-maltodextrin hydrogel
- Glucose-maltodextrin ingestion (Active Comparator): Ingestion of glucose and maltodextrin (glucose polymers) at a rate of 90 g carbohydrate per hour during two hours of treadmill running at 60%VO2peak.
  Interventions: Dietary Supplement: Glucose-maltodextrin

INTERVENTIONS:
Dietary Supplement: Fructose-maltodextrin — Fructose plus maltodextrin in a ratio of 1:1.4, diluted in water to produce a 16% carbohydrate solution.
  Arms: Fructose-maltodextrin ingestion
Dietary Supplement: Fructose-maltodextrin hydrogel — Fructose plus maltodextrin in a ratio of 1:1.4, encapsulated in an alginate-pectin hydrogel diluted in water to produce a 16% carbohydrate solution.
  Arms: Fructose-maltodextrin hydrogel ingestion
Dietary Supplement: Glucose-maltodextrin — Glucose plus maltodextrin in a ratio of 1:1.4, diluted in water to produce a 16% carbohydrate solution.
  Arms: Glucose-maltodextrin ingestion

SUMMARY:
The aim of this study is to characterise exogenous carbohydrate oxidation rates during exercise, when ingesting glucose (polymers) only, compared to glucose-fructose mixtures, and glucose-fructose mixtures ingested in hydrogel form.

ELIGIBILITY:
Inclusion Criteria:

* Maximal oxygen consumption > 50 ml.kg-1.min-1
* > 1 year training in endurance running or triathlon
* No current injury or injury within the last three months
* No history of cardiac or metabolic disease such as coronary heart disease or diabetes
* No current or history of gastrointestinal issues
* Successful completion of the physical activity readiness questionnaire (PAR-Q)

Exclusion Criteria:

* Female
* Untrained in endurance running
* Current injury or injury within the past three months
* History of cardiac or metabolic disease such as coronary heart disease or diabetes
* History of or current gastrointestinal issues such as irritable bowel syndrome
* Unable to replicate diet and training for 3 and 5 days respectively prior to each experimental visit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-10-14 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Peak exogenous carbohydrate oxidation rate | 120 minutes
  Peak exogenous carbohydrate oxidation rate during 120 min of treadmill running. Measured using isotope ratio mass spectrometry and reported in grams per minute

SECONDARY OUTCOMES:
Total carbohydrate oxidation | 120 minutes
  Total carbohydrate oxidation during 120 min of treadmill running. Measured using indirect calorimetry and reported in grams.
Ratings of gastrointestinal discomfort | 120 minutes
  Subjective ratings of gastrointestinal discomfort during 120 min of treadmill running. Measured using a 9-item questionnaire on a scale of 1 to 7, where 1 = No discomfort at all and 7 = very severe discomfort.
  Items: Stomach; Heartburn; Acid reflux; Nausea; Rumbling; Bloated; Burping; Passing gas; Bowel movement.
Total fat oxidation | 120 minutes
  Total fat oxidation during 120 min of treadmill running. Measured using indirect calorimetry and reported in grams.
Plasma insulin concentrations | 120 minutes
  Plasma insulin concentrations during 120 min of treadmill running. Measured using enzyme-linked immunosorbent assay and reported in pmol/L.
Plasma glucose concentrations | 120 minutes
  Plasma lactate concentrations during 120 min of treadmill running. Measured using colourimetric assay and reported in mmol/L.
Plasma lactate concentrations | 120 minutes
  Plasma lactate concentrations during 120 min of treadmill running. Measured using colourimetric assay and reported in mmol/L.
Plasma non-esterified fatty acid concentrations | 120 minutes
  Plasma insulin concentrations during 120 min of treadmill running. Measured using colourimetric assay and reported in umol/L.
Ratings of perceived exertion | 120 minutes
  Subjective ratings of perceived exertion using the Borg scale (1982) during 120 min of treadmill running. Measured on a scale of 6 to 20, where 6 = no exertion at all, and 20 = maximal exertion.
Heart rate | 120 minutes
  Heart rate during treadmill running measured by telemetry and reported in beats per minute.
Rate of oxygen consumption | 120 minutes
  Rate of oxygen consumption during 120 min of treadmill running. Measured using indirect calorimetry and reported in litres per minute.
Rate of carbon dioxide production | 120 minutes
  Rate of carbon dioxide production during 120 min of treadmill running. Measured using indirect calorimetry and reported in litres per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom